CLINICAL TRIAL: NCT03747341
Title: A Study Examining the Pharmacodynamics Interaction Between Buprenorphine and Fentanyl
Brief Title: Buprenorphine-Fentanyl Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: INDV-6000-101; 2017-004858-42 (EudraCT Number); CHDR1754 (Other: Centre for Human Drug Research)
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Opioid Use
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: Part A is a 3 period study in approximately 18 healthy subjects. Subjects will be randomized in a 1:1 ratio to 2 treatment sequences determined by the order in which they receive buprenorphine or placebo (periods 1 and 2). An optional open-label Period 3 may be conducted in which subjects will receive buprenorphine only.
  Part B is an open label study of approximately 8 opioid tolerant patients. All will undergo a washout of their own opioids which will be replaced with oral oxycodone and continue at stable doses from at least 48 hours prior to Period 1 to the end of Period 2. All will receive placebo plus fentanyl during Period 1 and buprenorphine plus fentanyl during Period 2.
Who Masked: Participant
Masking Description: Participants will be blinded to treatment with buprenorphine or placebo during Periods 1 and 2 in Part A only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part A (Healthy Participants): Placebo-Buprenorphine Low (Experimental): Three treatment periods consisting of 3 days each of investigational treatment
  * 1=placebo + fentanyl,
  * 2=low dose buprenorphine + fentanyl,
  * 3 (optional)=low dose buprenorphine only
  Fentanyl was administered as a bolus over 90 seconds in escalating doses of 0.075, 0.15, 0.25 and 0.35 mg/70 kg.
  Each dosing period was followed by 10-17 days of washout.
  Interventions: Drug: Buprenorphine Injectable Solution - Part A; Drug: Placebo - Parts A + B; Drug: Fentanyl - Part A; Drug: Ondansetron - Parts A + B
- Part A (Healthy Participants): Placebo-Buprenorphine High (Experimental): Three treatment periods consisting of 3 days each of investigational treatment
  * 1=placebo + fentanyl,
  * 2=high dose buprenorphine + fentanyl,
  * 3 (optional)=high dose buprenorphine only
  Fentanyl was administered as a bolus over 90 seconds in escalating doses of 0.075, 0.15, 0.25 and 0.35 mg/70 kg.
  Each dosing period was followed by 10-17 days of washout.
  Interventions: Drug: Buprenorphine Injectable Solution - Part A; Drug: Placebo - Parts A + B; Drug: Fentanyl - Part A; Drug: Ondansetron - Parts A + B
- Part A (Healthy Participants): Buprenorphine Low-Placebo (Experimental): Three treatment periods consisting of 3 days each of investigational treatment
  * 1=low dose buprenorphine + fentanyl,
  * 2=placebo + fentanyl,
  * 3 (optional)=low dose buprenorphine only
  Fentanyl was administered as a bolus over 90 seconds in escalating doses of 0.075, 0.15, 0.25 and 0.35 mg/70 kg.
  Each dosing period was followed by 10-17 days of washout.
  Interventions: Drug: Buprenorphine Injectable Solution - Part A; Drug: Placebo - Parts A + B; Drug: Fentanyl - Part A; Drug: Ondansetron - Parts A + B
- Part A (Healthy Participants): Buprenorphine High-Placebo (Experimental): Three treatment periods consisting of 3 days each of investigational treatment
  * 1=high dose buprenorphine + fentanyl,
  * 2=placebo + fentanyl,
  * 3 (optional)=high dose buprenorphine only
  Fentanyl was administered as a bolus over 90 seconds in escalating doses of 0.075, 0.15, 0.25 and 0.35 mg/70 kg.
  Each dosing period was followed by 10-17 days of washout.
  Interventions: Drug: Buprenorphine Injectable Solution - Part A; Drug: Placebo - Parts A + B; Drug: Fentanyl - Part A; Drug: Ondansetron - Parts A + B
- Part B (Opioid-Tolerant): Placebo-Buprenorphine Low (Experimental): Opioid-tolerant participants in Part B undergo a washout of their own opioids during which these were replaced with oral oxycodone, and continue at stable doses of oxycodone from at least 48 hours before Period 1 to the end of Period 2.
  Two treatment periods:
  * 1=placebo (Day 1),
  * 2=low dose buprenorphine + fentanyl (Day 3)
  Fentanyl was administered as a bolus over 90 seconds in escalating doses of 0.25, 0.35, 0.5 and 0.7 mg/70 kg.
  Interventions: Drug: Placebo - Parts A + B; Drug: Ondansetron - Parts A + B; Drug: Buprenorphine Injectable Solution - Part B; Drug: Fentanyl - Part B; Drug: Oxycodone - Part B
- Part B (Opioid-Tolerant): Placebo-Buprenorphine Mid (Experimental): Opioid-tolerant participants in Part B undergo a washout of their own opioids during which these were replaced with oral oxycodone, and continue at stable doses of oxycodone from at least 48 hours before Period 1 to the end of Period 2.
  Two treatment periods:
  * 1=placebo (Day 1),
  * 2=mid dose buprenorphine + fentanyl (Day 3)
  Fentanyl was administered as a bolus over 90 seconds in escalating doses of 0.25, 0.35, 0.5 and 0.7 mg/70 kg.
  Interventions: Drug: Placebo - Parts A + B; Drug: Ondansetron - Parts A + B; Drug: Buprenorphine Injectable Solution - Part B; Drug: Fentanyl - Part B; Drug: Oxycodone - Part B
- Part B (Opioid-Tolerant): Placebo-Buprenorphine High (Experimental): Opioid-tolerant participants in Part B undergo a washout of their own opioids during which these were replaced with oral oxycodone, and continue at stable doses of oxycodone from at least 48 hours before Period 1 to the end of Period 2.
  Two treatment periods:
  * 1=placebo (Day 1),
  * 2=high dose buprenorphine + fentanyl (Day 3)
  Fentanyl was administered as a bolus over 90 seconds in escalating doses of 0.25, 0.35, 0.5 and 0.7 mg/70 kg.
  Interventions: Drug: Placebo - Parts A + B; Drug: Ondansetron - Parts A + B; Drug: Buprenorphine Injectable Solution - Part B; Drug: Fentanyl - Part B; Drug: Oxycodone - Part B

INTERVENTIONS:
Drug: Buprenorphine Injectable Solution - Part A — Buprenorphine intravenous (IV) injection given as a primed-continuous infusion.
  Low Dose: initial bolus (0.05 mg/70 kg) administered over 15 minutes and infusion continued (0.02 mg/70 kg/hour infusion rate) to complete 360 minutes of administration targeting 0.2 ng/ml.
  High Dose: initial bolus (0.125 mg/70 kg) administered over 15 minutes and infusion continued (0.05 mg/70 kg/hour infusion rate) to complete 360 minutes of administration targeting 0.5 ng/ml.
  Administration of buprenorphine was flexible and infusion rates were selected to target approximately 25 to 50% respiratory depression.
  Other Names: TEMGESIC®
  Arms: Part A (Healthy Participants): Buprenorphine High-Placebo; Part A (Healthy Participants): Buprenorphine Low-Placebo; Part A (Healthy Participants): Placebo-Buprenorphine High; Part A (Healthy Participants): Placebo-Buprenorphine Low
Drug: Placebo - Parts A + B — 0.9% normal saline for IV administration was used as placebo matching the buprenorphine formulation and administration.
Drug: Fentanyl - Part A — Participant received up to four fentanyl doses: 0.075, 0.15, 0.25, and 0.35 mg/70 kg in Periods 1 and 2. Fentanyl boluses were administered over 90 seconds by dose escalation +2hr, +3hr, +4hr and +5hr after starting administration of buprenorphine/ placebo. Administration of fentanyl was flexible and bolus doses were selected to elicit moderate to more severe respiratory depression with apnoea ≥20 seconds.
  Arms: Part A (Healthy Participants): Buprenorphine High-Placebo; Part A (Healthy Participants): Buprenorphine Low-Placebo; Part A (Healthy Participants): Placebo-Buprenorphine High; Part A (Healthy Participants): Placebo-Buprenorphine Low
Drug: Ondansetron - Parts A + B — A non-investigational intervention administered as an infusion prior to investigation intervention. 4 mg of ondansetron was administered to manage the expected gastrointestinal side effect (nausea, vomiting) to buprenorphine.
Drug: Buprenorphine Injectable Solution - Part B — Buprenorphine intravenous (IV) injection given as a primed-continuous infusion.
  Low Dose: initial bolus (0.25 mg/70 kg) administered over 15 minutes and infusion continued (0.1 mg/70 kg/hour infusion rate) to complete 360 minutes of administration targeting 1 ng/ml.
  Mid Dose: initial bolus (0.5 mg/70 kg) administered over 15 minutes and infusion continued (0.2 mg/70 kg/hour infusion rate) to complete 360 minutes of administration targeting 2 ng/ml.
  High Dose: initial bolus (1.25 mg/70 kg) administered over 15 minutes and infusion continued (0.5 mg/70 kg/hour infusion rate) to complete 360 minutes of administration targeting 5 ng/ml.
  Other Names: TEMGESIC®
  Arms: Part B (Opioid-Tolerant): Placebo-Buprenorphine High; Part B (Opioid-Tolerant): Placebo-Buprenorphine Low; Part B (Opioid-Tolerant): Placebo-Buprenorphine Mid
Drug: Fentanyl - Part B — Participant received up to four fentanyl doses: 0.25, 0.35, 0.5, and 0.7 mg/70 kg in Periods 1 and 2.
  Fentanyl boluses were administered over 90 seconds by dose escalation +2hr, +3hr, +4hr and +5hr after starting administration of buprenorphine/ placebo.
  Arms: Part B (Opioid-Tolerant): Placebo-Buprenorphine High; Part B (Opioid-Tolerant): Placebo-Buprenorphine Low; Part B (Opioid-Tolerant): Placebo-Buprenorphine Mid
Drug: Oxycodone - Part B — All opioid-tolerant participants in Part B were transitioned to oral oxycodone at least 48 hours before Period 1 to ensure washout of the participants' regular opioids and a stable dose of oxycodone with an adequate bridging schedule reached. Oxycodone is a non-investigational intervention.
  Arms: Part B (Opioid-Tolerant): Placebo-Buprenorphine High; Part B (Opioid-Tolerant): Placebo-Buprenorphine Low; Part B (Opioid-Tolerant): Placebo-Buprenorphine Mid

SUMMARY:
An increase in overdose deaths has been attributed to widespread access to fentanyl and carfentanyl. The study is designed to determine if buprenorphine can change the respiratory depression response to intravenous (IV) fentanyl.

DETAILED DESCRIPTION:
The study will be performed in 2 parts. Part A is a 3-period study; the first 2 periods have a single-blind, placebo-controlled, cross-over design, where subjects will be randomized in a 1:1 ratio to 2 treatment sequences determined by the order in which they receive buprenorphine or matching placebo. Period 3 is an open-label design where the same subjects will receive buprenorphine only. This period is optional, and will include approximately 6 subjects.

Part B is an open-label study in opioid tolerant patients. All will receive placebo plus fentanyl in Period 1 to permit dose escalation to full respiratory effects of fentanyl before assessing the interaction with buprenorphine. Subjects will receive buprenorphine plus fentanyl during Period 2 to assess the interaction with buprenorphine.

To study ventilation, the dynamic end-tidal forcing technique will be used. This technique enables the Investigator to force end-tidal partial pressure of carbon dioxide and end-tidal partial pressure of oxygen to follow a specific pattern in time. Subjects with a procedure-related adverse event (AE) will be treated according to established ventilatory support and opioid reversal protocols.

ELIGIBILITY:
Inclusion Criteria:

* Part A-Healthy Subjects:

  1. Signed the informed consent form (ICF) and able to comply with study requirements and restrictions
  2. Age 18- 45, inclusive years for this part
  3. Women of childbearing potential must have a negative serum pregnancy test prior to enrolment and must agree to use a medically acceptable means of contraception through at least 3 months after last dose of study drug
  4. Body Mass Index (BMI) 18-30 kg/m^2, inclusive
  5. Healthy as defined by the Investigator
  6. No history of substance use disorder
  7. No current use of any central nervous system (CNS) depressants
* Part B-Opioid-tolerant patients

  1. Signed the ICF and able to comply with study requirements and restrictions
  2. Age 18 - 55 years inclusive
  3. Same as #3 above
  4. BMI 18-32 kg/m^2
  5. Opioid tolerant patients administered opioids at daily doses greater than or equal to 90 mg oral morphine equivalents
  6. Stable as defined by the Investigator
  7. No current use of any CNS depressants, besides opioids, for 5 half-lives of the product before first study drug administration

Exclusion Criteria:

Part A

1. History of risk factors of Torsades de Pointes or an electrocardiogram (ECG) demonstrating a Fridericia's corrected QT interval (QTcF) > 450 msec in males and QTcF > 470 msec in females at screening;
2. Currently meet the criteria for diagnosis of substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria on any substance;
3. Any other active medical condition, organ disease or concurrent medication or treatment that may either compromise subject safety or interfere with study endpoints;
4. Current smokers and those who have smoked within the last 6 months;
5. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 6 months;
6. Consume, on average, > 20 units/week of alcohol in men and > 13 units/week of alcohol in women; (1 unit = 1 glass (250 mL) beer, 125 mL glass of wine or 25 mL of 40% spirit);
7. Previous treatment with any prescribed medications (including all types of vaccines) or over-the-counter (OTC) medications within 14 days or 5 half-lives (whichever is longer) prior to first study treatment administration;
8. Previous or current treatment with opioid agonist, partial agonist, or antagonist treatment within 30 days prior to the first study drug administration;
9. Require ongoing prescription or OTC medications that are clinically relevant cytochrome (CYP) P450 3A4 or CYP P450 2C8 inducers or inhibitors;
10. Significant traumatic injury, major surgery, or open biopsy within the prior 4 weeks of informed consent;
11. History of suicidal ideation within 30 days prior to informed consent or history of a suicide attempt in the 6 months prior to informed consent;
12. Measured systolic blood pressure greater than 160 or less than 95 mmHg or diastolic pressure greater than 95 mmHg prior to Day 1;
13. History or presence of allergic response to buprenorphine or fentanyl;
14. Subjects who have demonstrated allergic reactions which, in the opinion of the Investigator and sponsor, interfere with their ability to participate in the trial;
15. Estimated glomerular filtration rate <60 mL/min as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation;
16. Anaemia at screening or donation of > 250 mL of blood or plasma within the last 3 months;
17. Positive serology tests for human immunodeficiency virus (HIV), hepatitis B (HBsAg), or hepatitis C (HepC);
18. Aspartate transaminase (AST) or alanine transaminase (ALT) levels >1.5 times the upper limit of normal at screening;
19. Treatment with another investigational drug within 3 months prior to dosing or having participated in more than 4 investigational drug studies within 1 year prior to screening;
20. Site staff or subjects affiliated with, or a family member of, site staff directly involved in the study.

Part B

1. Same as Part A #1
2. Currently meet the criteria for diagnosis of moderate or severe substance use disorder according to the DSM-5 criteria on any substances other than opioids, caffeine or nicotine;
3. Same as Part A #3;
4. Smoking of >10 cigarettes/day or equivalent and not able to abstain from smoking cigarettes during each dose administration day;
5. Consume, on average, >27 units/week of alcohol in men and >20 units/week of alcohol in women;
6. Use of buprenorphine within 10 days of the first study drug administration;
7. Require ongoing prescription or OTC medications that are clinically relevant CYP P450 3A4 or CYP P450 2C8 inducers or inhibitors;
8. Significant traumatic injury, major surgery, or open biopsy within the prior 4 weeks of informed consent;
9. History of suicidal ideation within 30 days prior to informed consent or history of a suicide attempt in the 6 months prior to informed consent;
10. Measured systolic blood pressure greater than 160 or less than 95 mmHg or diastolic pressure greater than 95 mmHg prior to Day 1;
11. History or presence of allergic response to buprenorphine or fentanyl;
12. Opioid-tolerant patients who have demonstrated allergic reactions which, in the opinion of the Investigator and sponsor, interfere with their ability to participate in the trial;
13. Same as Part A #15
14. Same as Part A #16
15. Same as Part A #17
16. Same as Part A #18
17. Same as Part A #19
18. Same as Part A #20

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — For Part A, at least 5 subjects of each sex will be included in the population. For Part B, at least 3 patients of each sex will be included
Enrollment: 22 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Changes in peak ventilatory depression will be measured. | 6 hours (during study drug infusion)
  Peak ventilatory depression (change in minute ventilation) will be calculated based on a 1-minute average of the ventilation data of each individual subject/patient. For buprenorphine or placebo, absolute changes and percentage changes are calculated from the baseline value. For fentanyl, absolute changes and percentage changes for each bolus are calculated from the baseline value and from the pre-fentanyl baseline value immediately before the first fentanyl bolus

SECONDARY OUTCOMES:
Number (percentage) of subjects who experience apnoea for each fentanyl dose during the placebo treatment vs. the buprenorphine treatment | 6 hours
  Apnoea is defined as a 20-second pause in respiration. If apnoea is observed at any fentanyl dose, the subject will be classified as "experienced apnoea" for that dose and any higher dose planned will be withheld
Number (percentage) of subjects who require stimulation for breathing for each fentanyl dose during the placebo treatment vs. the buprenorphine treatment. | 6 hours
  If a subject required stimulation for breathing at a fentanyl dose and the next higher dose was withheld, the subject will be classified as requiring breath stimulation for all withheld doses

CONTACTS AND LOCATIONS:
Overall Officials: Geert J Groeneveld, Principal Investigator — Center for Human Drug Research
Locations (1):
- Center for Human Drug Research, Leiden, The Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olofsen E, Algera MH, Moss L, Dobbins RL, Groeneveld GJ, van Velzen M, Niesters M, Dahan A, Laffont CM. Modeling buprenorphine reduction of fentanyl-induced respiratory depression. JCI Insight. 2022 May 9;7(9):e156973. doi: 10.1172/jci.insight.156973. PMID 35316224
- [Result] Moss LM, Algera MH, Dobbins R, Gray F, Strafford S, Heath A, van Velzen M, Heuberger JAAC, Niesters M, Olofsen E, Laffont CM, Dahan A, Groeneveld GJ. Effect of sustained high buprenorphine plasma concentrations on fentanyl-induced respiratory depression: A placebo-controlled crossover study in healthy volunteers and opioid-tolerant patients. PLoS One. 2022 Jan 27;17(1):e0256752. doi: 10.1371/journal.pone.0256752. eCollection 2022. PMID 35085249